CLINICAL TRIAL: NCT07002424
Title: A Protocol for a Pilot and Feasibility Randomised Controlled Trial of an Online Cancer Bereavement Group.
Brief Title: Feasibility and Outcomes of Therapist-led Online Cancer Bereavement Groups
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Project 0183
Record Dates: First submitted 2025-05-12; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Waitlist Control; Intervention (Training) Condition
Keywords: Online Bereavement Group; Cancer Loss; Therapist-Led

STUDY DESIGN:
Intervention Model Description: It will use a longitudinal pilot and feasibility methodology to evaluate a randomised controlled trial (RCT) design and its suitability for a further full-scale RCT. The study will include two parallel conditions: non-waitlist (online bereavement group), and a wait-list control condition.
  Four groups are planned: Two whereby participants will be randomised to waitlist (WL) accessing the intervention after a delay and two with participants randomised to non-waitlist (non-WL), accessing the intervention immediately. Both groups will run simultaneously (twice a week, over 8 sessions covering a period of 12 weeks) but the WL groups will run parallel to the non-WL groups, three months later. Assessments will be conducted at baseline and post each session and post-intervention 3 months later.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants randomised to non-waitlist, accessing the online bereavement group intervention immediately
  Interventions: Behavioral: Therapeutic - Psychological
- Waitlist-Control Group (Other): participants randomised to waitlist-control accessing the online bereavement group intervention after a delay (three months later) immediate group
  Interventions: Behavioral: Therapeutic - Psychological

INTERVENTIONS:
Behavioral: Therapeutic - Psychological — The intervention uses a transdiagnostic model that incorporates aspects of peer support, psychoeducation, trauma-informed cognitive behavioural therapy (CBT), Compassion focused therapy (CFT) models of distress. It also aligns itself to the Dual Processing Model of coping with bereavement (Stroebe & Schut, 2010) and Tonkin's model of grief (Tonkin, 1996).

SUMMARY:
Background: The loss of loved one to cancer brings unique difficulties that impact on the bereavement experience. Mixed support exists for the effectiveness of in-person group interventions for bereaved caregivers, with barriers to accessing support including perceived stigmatisation and geographical constraints. Online bereavement interventions offer an accessible and effective means of providing grief support to various populations at the individual and group level. Research supports the effectiveness of online groups for those bereaved by cancer, although most of these studies are peer-led as opposed to therapist-led. Despite a growing rationale for the use of online groups for bereavement, there is little empirical evidence for therapist led groups, or for those bereaved by cancer. Objectives: This paper describes the protocol for a pilot feasibility trial evaluating the feasibility, potential effectiveness and acceptability of delivering online therapy groups for those bereaved by cancer. Methods and analysis: It will use a longitudinal pilot and feasibility methodology to evaluate a randomised controlled trial (RCT) design and its suitability for a future definitive RCT. Participants: A total of 100 adults who have lost a loved one to cancer will be randomised to receive the intervention immediately or after a delay three months later. Interventions: An eight-session online therapeutic group intervention led over 12 weeks based on models of cognitive behavioural therapy, compassion focused therapy and coping with bereavement. Primary outcome measures: Cancer- bereaved adults' grief intensity, depression, anxiety, PTSD, self-compassion and social disconnection. Acceptability of the intervention will also be measured including what participants found most helpful or unhelpful about the groups and any adverse outcomes. Data collection will occur at baseline, intervention completion and at follow up, 3 months after intervention completion. Results: The feasibility of trial procedures and the effect of the intervention on the outcomes will be tested,. Conclusions: At intervention completion, it is hoped that participants will show reductions across all outcomes measures with improvements remaining at follow up, compared to the waitlist-control group, warranting the need for a full-scale RCT to establish efficacy. Trial registration (intended registry): Protocol version: 1 (No amendments currently), Issued:

DETAILED DESCRIPTION:
The loss of a loved one to cancer brings unique difficulties that impact the bereavement experience. Mixed evidence exists for the effectiveness of in-person group interventions for bereaved caregivers, with barriers to access including perceived stigmatisation and geographical constraints. Online bereavement interventions offer an accessible, destigmatising and effective means of providing grief support to various populations at the individual and group level. Research supports the effectiveness for online groups for those bereaved by cancer, although most of these studies are peer-led as opposed to therapist-led. Despite a growing rationale for the use of online groups for bereavement, there is little (if any) empirical evidence for therapist led groups, or for those bereaved by cancer.

A group bereavement therapy programme was developed by the Loss Foundation, a national cancer bereavement charity, who initiated the project. It will explore the impact of an eight-session therapeutic group intervention led over 12 weeks on cancer- bereaved adults' grief intensity, depression, anxiety, PTSD, self-compassion and social disconnection. Previous research within the Loss Foundation has demonstrated the effectiveness of an in-person cancer bereavement therapeutic group using a transdiagnostic model (Jerome et al., 2018). In this study, it was found that grief intensity and symptoms of posttraumatic stress disorder (PTSD), depression, and anxiety were reduced postintervention, and self-compassion increased. At follow-up, improvement remained for grief, PTSD, and depression. This intervention has been adapted and carried out several times from previous research, including methodological changes such as randomisation to a waitlist control and collection of weekly data. For example, previous research within The Loss Foundation explored the effectiveness of the in-person cancer bereavement therapeutic group compared to waitlist control with findings showing a reduction in grief intensity and increased self-compassion.

As this is the first online therapeutic bereavement group for those bereaved by cancer, this study offers a unique contribution to the literature, addressing a critical gap in the literature on evidence-based therapist led internet interventions for cancer bereaved adults. The intention is to ascertain the feasibility, acceptability and changes in self-report measures of the online version of the adapted group bereavement therapy programme for cancer. This feasibility pilot study will evaluate a randomised controlled trial (RCT) design to explore its suitability for a further full-scale RCT. Outcomes will be assessed by comparing intervention and wait-list control groups at baseline, post each session and postintervention 3 months later in terms of the following primary outcomes: grief intensity, depression, anxiety, PTSD, self-compassion and social disconnection.

Aims and objectives

1. The primary aim is to evaluate the feasibility and acceptability of delivering online bereavement group for cancer loss. This refers to feasibility to recruit, retain, randomise and acceptability as tracking participant satisfaction and any adverse outcomes.
2. The secondary aim is to explore the preliminary effectiveness by examining whether the online bereavement group intervention leads to improvements on various outcomes, compared to the waitlist control.

The investigators' hypotheses are informed by the results of previous research within The Loss Foundation, and previous literature suggesting that online groups may be similarly effective. In regard to the secondary aim of exploring preliminary effectiveness of the study, the investigators hypothesised that grief intensity and PTSD symptoms, depression, and anxiety will be reduced postintervention, and self-compassion will be increased, showing improvement from baseline, compared to the waitlist control. Further, the investigators hypothesise that at follow-up, improvement will be maintained for grief intensity, PTSD symptoms and depression.

ELIGIBILITY:
Inclusion Criteria:

* (1) Adults (aged 18 or over) who are bereaved by cancer, for example losing a partner, family member or friend
* (2) The time since death must have been more than 6 months, so as not to interfere with a natural recovery process (Henk Schut & Stroebe, 2010)
* (3) Self-referral to The Loss Foundation or via a related organisation
* (4) Have the means to access the therapeutic group online
* (5) Participants consent to attending the intervention with the risk of a delay (e.g. by being randomised to the waitlist or non-waitlist group).

Exclusion Criteria:

1. Adults at high risk to themselves or others in regard to suicide and/or self-harm
2. Significant substance or alcohol misuse which would interfere with participants' ability to take part in the research
3. Cannot be involved in other therapy at the same time elsewhere.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Mood Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001) | Baseline (1 week pre-group) Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  is a 9-item self-report questionnaire that measures the severity of depressive symptoms. Kroenke et al. (2001) reported that the measure has strong psychometric properties: the internal consistency was 0.89 and test-retest reliability between patient self-report and mental health professional administering the measure telephonically 48 hours later was 0.84. The measure also has good convergent validity (r=0.73) with the mental health subscale of the Short- Form General Health Surv. The PHQ-9 has not been validated with bereaved populations.
Generalized Anxiety Disorder-7 (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) | Baseline (1 week pre-group) Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  is a 7-item self-report questionnaire that measures the severity of anxiety symptoms. Spitzer et al., (2006) reported that the measure has strong psychometric properties: the internal consistency was 0.92 and test-retest reliability was 0.83 over a period of a week. The measure has strong convergent validity with the Beck Anxiety Inventory (r=0.72) and the anxiety sub-scale of the Symptom Checklist-90 (r=0.74). The GAD-7 has not been validated with bereaved populations.
Prolonged Grief Disorder (PG - 13) (Prigerson et al., 2008) | Baseline (1 week pre-group) Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  13-item self-report measure that examines three facets of prolonged grief disorder: feelings, thoughts and actions, occurring over the past month. The measure has strong psychometric properties. For example, Ashouri et al., (2024) found that this measure demonstrated good internal consistency (omega coefficient of 0.93), and test-retest reliability with an interval of 6 weeks being 0.89. The PG-13 was shown to be a reliable scale for the assessment of individuals at risk for developing PGD with high scores on internal consistency in bereaved Swedish parents (Pohlkamp et al., 2018). However, these properties have been validated with a few studies.
PTSD Checklist for DSM-5 | Baseline (1 week pre-group) Session 4(week 4) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  is a 20-item self-report questionnaire that assesses symptoms of PTSD. Blevins et al., (2015) reported that the measure has strong psychometric properties: when tested with trauma-exposed undergraduate students, the internal consistency was 0.94 and the test-retest reliability was 0.82 over a period of a week. There appears to be no validation of the PCL-5 targeting traumatically bereaved individuals.
The Helpful Aspects of Therapy (HAT; Llewelyn, 1988) | Session 1 (Week 1) Session 2 (week 2) Session 3 (week 3) Session 4 (week 4) Session 5 (week 6) Session 6 (week 8) Session 7 (week 10) Session 8 (week 12)
  is a post-session self - report questionnaire that asks about perceptions of key change processes in therapy. It is partly qualitative and captures perceptions of helpful and unhelpful aspects of the previous session. It is beyond the scope of this present study to analyse the qualitative data, however this measure provides valuable feedback, which the facilitators can be aware of and address if appropriate.
  Researchers will aim to foster trusting relationships to help the participants to feel engaged in the research process. Participants will be given opportunities to share their thoughts and reflections during the group to facilitate engagement with the content.
The Self-Compassion Scale (SCS; Neff, 2003) | Baseline (1 week pre-group) Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  is a 26-item self-report questionnaire that measures self-compassion. Raes et al. (2011) reported that the measure has strong psychometric properties: the internal consistency was 0.85 and the test-retest reliability over a period of five months was 0.71. The total score of the SCS-SF correlates highly (r=0.98) with the longer 26-item Self-Compassion Scale. Construct validity of the SCS-SF has not been tested but the long version of the SCS was negatively correlated (r=-0.65) with the self-criticism subscale of the Depressive Experiences Questionnaire. The SCS-SF has not been validated with bereaved populations.
Oxford Grief-Social Disconnection Scale (OG-SD; Smith et al., 2020) | Baseline (1 week pre-group) Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  is a 15-item scale developed from interviews with bereaved individuals. Smith et al., (2020) indicate that internal consistency for the total OG-SD and its subscales were good or excellent (Cronbach alpha 0.80). The OG-SD showed a good 7-day-retest reliability across the total and subscales, indicating a temporally stable assessment of perceived social disconnection (test-retest 0.94). However, although overall the OG-SD was deemed stable over time, other two subscales may be less stable over time. The test-retest sample was also relatively small, which means that it is possible that large effects may have been caused within a few individuals.

SECONDARY OUTCOMES:
Demographic Information- Name | Baseline (1 week pre-group) Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information- Address | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information - Age | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information- Gender | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information- Ethnicity | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. The data securely stored and we have ethical approval to capture special category data for example ethnicity.
Demographic Information- Marital status | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information- Highest level qualification | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information- Employment | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information- Psychological treatment since bereavement | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Demographic Information - Gender of deceased | Baseline (1 week pre-group)
  As part of group therapeutic interventions, The Loss Foundation routinely collects outcome measures and demographic information to evaluate the effectiveness of its services. For therapy groups, the data securely stored.
Bereavement characteristics: Length of relationship with deceased | Baseline (1 week pre-group)
  Bereavement characteristics are also routinely collected by the Loss Foundation:
Bereavement characteristics -Time since death | Baseline (1 week pre-group)
Bereavement characteristics - Relationship with deceased | Baseline (1 week pre-group)
Bereavement characteristics - Co-habiting with deceased prior to death | Baseline (1 week pre-group)
Bereavement characteristics - Contact with deceased prior to death | Baseline (1 week pre-group)
- Bereavement characteristics Frequency of seeing deceased in 3 months preceding death | Baseline (1 week pre-group)
Bereavement characteristics Present at the death, | Baseline (1 week pre-group)
Bereavement characteristics - death of other loved ones in past 3 years. | Baseline (1 week pre-group)
Recruitment and uptake-Source of referral to the study | Baseline (1 week pre-group)
Recruitment and uptake- number consenting to participate | Baseline (1 week pre-group)
Recruitment and uptake- those eligible/willing to be randomised. | Baseline (1 week pre-group)
Adherence and attrition- A record of participation completion of outcome measurements | Baseline (1 week pre-group) Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12) Follow up (3 months post-group) WL: Additional follow up (3months post Baseline)
  Participants will also be prompted by 2-3 reminder emails to complete the outcome measures post each session
Adherence and attrition- Attendance | Session 1(Week 1) Session 2(week 2) Session 3(week 3) Session 4(week 4) Session 5(week 6) Session 6(week 8) Session 7(week 10) Session 8(week 12)
  Captured by the zoom meeting report stored on TLF secure server. We let them know as part of the screening process that the programme builds on material session by session and therefore full attendance is required for maximum benefit.
  Participants will be asked to complete homework tasks to provide participants with the opportunity to practice and apply the skills and ideas discussed in the sessions as well as develop a sense of self-responsibility. A follow up email will be sent after each session to remind of their home task and self-care.
Acceptability - Intervention | Session 8(week 12- 1 week post-group), Follow up 2 (3 months post-group).
  Satisfaction with therapy group (Likert scale)
Acceptability- Adverse cirumstances | Session 8(week 12- 1 week post-group), Follow up 2 (3 months post-group).
  Feeling supported in distress both during an outside sessions (Likert scale)
Acceptability- Intervention Content | Session 8(week 12- 1 week post-group), Follow up 2 (3 months post-group).
  Content preference (open ended)
Acceptability- Online modality | Session 8(week 12- 1 week post-group), Follow up 2 (3 months post-group).
  Experience of online modality of group as opposed to in person (Likert scale)
Acceptability- Facilitator effectiveness | Session 8(week 12- 1 week post-group), Follow up 2 (3 months post-group).
  Facilitator effectiveness in. Likert scale of: Created a safe and supportive space, Treated group members with respect and empathy, Kept the group on track while allowing flexibility, Managed difficult group dynamics effectively, Delivered clear explanations that helped me to learn about my grief and how to manage it
Acceptability- Group size | Session 8(week 12- 1 week post-group), Follow up 2 (3 months post-group).
  Acceptability- size of the group (Likert scale) impacting on engagement, connection with others, learning effectiveness, comfort expressing self

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Cole, Clinical Psychologist, Principal Investigator — University College, London
Locations (1):
- The Loss Foundation (Charity), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We hope to submit the paper and systematic review for publication in a peer-reviewed journals (e.g. The Journal of Loss and Trauma). Reports will not reveal the identity of anyone who took part. The consent form outlines to participants that their information provided for this study will be published as a report and they will be asked if they would like to receive a copy of it.
  Data management and monitoring has been registered and approved by the Data Protection Office (reference No Z6364106/2024/11/103 cancer research) in line with UCL's Data Protection Policy. All anonymised data generated or analysed during this study are included in this published article [and its supplementary information files].

REFERENCES:
- [Background] Jerome H, Smith KV, Shaw EJ, Szydlowski S, Barker C, Pistrang N, Thompson EH. Effectiveness of a Cancer Bereavement Therapeutic Group. J Loss Trauma. 2019 Jan 7;23(7):574-587. doi: 10.1080/15325024.2018.1518772. PMID 30983910